CLINICAL TRIAL: NCT05335577
Title: Concentrations of Urinary Claudin-2, Caveolin-1, and Epidermal Growth Factor (EGF) as the Prototypes of Non-Invasive Biomarkers in the Diagnosis of Necrotizing Enterocolitis in Preterm Neonates
Brief Title: Role of Urinary Claudin-2, Caveolin-1, and EGF as Diagnostic Biomarkers of Necrotizing Enterocolitis in Preterm Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Brawijaya (Other)
Responsible Party: Principal Investigator, Brigitta Ida Resita Vebrianti Corebima, dr. Brigitta Ida Resita Vebrianti Corebima, Sp.A(K), M.Kes, M.D.(Paed), Neonatology Division, Department of Pediatrics, Faculty of Medicine, Saiful Anwar General Hospital-University of Brawijaya, University of Brawijaya
Other Study IDs: 400/011/K.3/302/2022
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Enterocolitis, Necrotizing; Infant, Premature
Keywords: Necrotizing enterocolitis; Preterm neonates; Claudin-2; Caveolin-1; Epidermal growth factor; Bell's Criteria
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — Biospecimen to be retained are urine with volume of 10 cc, feces with mass of ±40 mg, and serum with volume of 3 cc in EDTA vacutainer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preterm neonates with NEC: Preterm neonates with gestational age of 28-32 weeks and diagnosed with Necrotizing Enterocolitis based on Bell's modification criteria.
  Interventions: Diagnostic Test: Urinary Claudin-2; Diagnostic Test: Urinary Caveolin-1; Diagnostic Test: Urinary EGF
- Preterm neonates without NEC: Preterm neonates with gestational age of 28-32 weeks and without Necrotizing Enterocolitis based on Bell's modification criteria.
  Interventions: Diagnostic Test: Urinary Claudin-2; Diagnostic Test: Urinary Caveolin-1; Diagnostic Test: Urinary EGF
- Healthy term neonates: Term neonates with gestational age of 37-42 weeks without any comorbidities.
  Interventions: Diagnostic Test: Urinary Claudin-2; Diagnostic Test: Urinary Caveolin-1; Diagnostic Test: Urinary EGF

INTERVENTIONS:
Diagnostic Test: Urinary Claudin-2 — A sequential non-invasive urinary molecular profiling for protein, i.e. Claudin-2 as potential marker for enterocyte tight junction disruption, would be analyzed quantitatively with ELISA and then compared between groups to assess the optimum sensitivity and specificity.
Diagnostic Test: Urinary Caveolin-1 — A sequential non-invasive urinary molecular profiling for protein, i.e. Caveolin-1 as potential marker for enterocyte tight junction disruption, would be analyzed quantitatively with ELISA and then compared between groups to assess the optimum sensitivity and specificity.
Diagnostic Test: Urinary EGF — A sequential non-invasive urinary molecular profiling for protein, i.e. epidermal growth factor (EGF) as potential marker for tight junction protective regulator, would be analyzed quantitatively with ELISA and then compared between groups to assess the optimum sensitivity.

SUMMARY:
Our study aims to determine the differences in the concentration of urinary claudin-2, caveolin-1, and epidermal growth factor (EGF) as non-invasive biomarkers in the diagnosis of Necrotizing Enterocolitis (NEC). We compare the concentration of urinary claudin-2, caveolin-1, and EGF between preterm neonates at risk of NEC and healthy term infants as the basis for determining NEC biomarkers with the most optimum sensitivity and specificity. This analytical observational study is based on biomolecular profiling with a prospective cohort design approach. The research subjects are a group of preterm neonates (gestational age of 28-34 weeks) who were admitted in Perinatology Unit, Department of Pediatrics, Saiful Anwar General Hospital, Malang and whom diagnosed with NEC using Bell's criteria and serum TGF-β levels. Subjects are selected by consecutive sampling and single-blind analysis was performed in the Laboratory of Bioscience and Biomedicine, Faculty of Medicine, University of Brawijaya.

During the research process, groups of preterm and term neonates would be observed and their clinical development followed. The collection of biologic samples would be taking 10 cc of urine and 40 mg of feces on day-5 (D5) and 7 (D7). The consecutive manner of urinary sampling was regarded to assess whether there was a time-related protein expression in the course of the NEC process. Faecal samples would be assessed for microbiota profile analysis described by the ratio of Proteobacteria: Firmicutes and Bacteroidetes to represent dysbiosis process in NEC. After 7 days, the subjects would be grouped into a group of preterm neonates with NEC, a group of healthy term neonates as a control, while a group of preterm infants at whom during the course of the study did not develop NEC, would be assigned to group of premature neonates without NEC.

Urinary protein concentrations from the three groups would then be analyzed and adjusted with normalized creatinine, so that the levels of these three proteins could be assessed quantitatively using the ELISA (Enzyme-Linked Immunosorbent Assay) method. The results would be compared with the microbiota profile as the golden standard for NEC cases. Through statistical tests, sensitivity, specificity and cut-off of selected protein levels would be assessed as diagnostic biomarkers of NEC.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is a multifactorial syndrome of acute intestinal ischemic necrosis which is one of the acute intestinal emergencies in neonates with high morbidity and mortality rates were higher in preterm. Inflammation and ischemia are the main pathogenesis of NEC. The diagnosis of NEC is established based on the demographic condition and clinical presentations, and further confirmed by the presence of pneumatosis intestinalis on plain abdominal radiographs. However, the clinical symptoms of NEC were often overlapped with other cases, especially diseases related to inflammation and sepsis, and the limitations of diagnostic methods both clinically and radiologically in identifying the early phase of NEC, make biomarker studies continue to be carried out to find diagnostic methods that would be able to predict, diagnose and differentiate NEC from non-NEC cases in a timely manner. Thus, a diagnostic method with high sensitivity and specificity is needed in cases of NEC in premature infants.

Several studies have shown that the immaturity of the gastrointestinal tract is related to the condition of the gastrointestinal cell barrier in infants who are susceptible to disintegration. The disruption in the expression of various proteins that make up the gastrointestinal tight junction in NEC, makes the tight junction protein component suspected to be a potential biomarker in the early phase of NEC. This is closely related to the presence of the inflammatory process of the NEC. Inflammatory conditions disrupt intestinal microcirculation, which results in the emergence of intestinal ischemia, and trigger the degradation of the tight junction components of the gastrointestinal tract through urine. This degradation process occurs in the early phase of the NEC disease course.

Several animal studies have shown that there is a correlation between abnormal expression of the proteins claudin-2, caveolin-1, and EGF and tight junction damage in NEC. Meanwhile, studies with a small number of neonates showed that the protein component is expressed in urine as a biomarker of tight junction damage in NEC and is independent of other inflammatory components, so that it is considered as a potential diagnostic biomarker in NEC cases.

This study aims to determine the differences in the expression of urinary claudin-2, caveolin-1, and EGF with NEC in preterm neonates at risk of NEC compared to healthy term infants as a basis for determining NEC biomarkers with optimum sensitivity and specificity, which then would be used as biomarker. The study was conducted using a cohort prospective method. The research subjects are a group of preterm neonates (gestational age of 28-34 weeks) who were admitted in Perinatology Unit, Department of Pediatrics, Saiful Anwar General Hospital, Malang and whom diagnosed with NEC using Bell's criteria and serum TGF-β levels obtained at Day-1 (D1). Subjects are selected by consecutive sampling and single-blind analysis was performed in the Laboratory of Bioscience and Biomedicine, Faculty of Medicine, University of Brawijaya.

During the research process, groups of preterm and term neonates would be observed and their clinical development followed. The collection of biologic samples would be taking 10 cc of urine and 40 mg of feces on day-5 (D5) and 7 (D7). The consecutive manner of urinary sampling was regarded to assess whether there was a time-related protein expression in the course of the NEC process. Faecal samples would be assessed for microbiota profile analysis described by the ratio of Proteobacteria: Firmicutes and Bacteroidetes to represent dysbiosis process in NEC. After 7 days, the subjects would be grouped into a group of preterm neonates with NEC, a group of healthy term neonates as a control, while a group of preterm infants at whom during the course of the study did not develop NEC, would be assigned to group of premature neonates without NEC.

Urinary protein concentrations from the three groups would then be analyzed and adjusted with normalized creatinine, so that the levels of these three proteins could be assessed quantitatively using the ELISA (Enzyme-Linked Immunosorbent Assay) method. The results would be compared with the microbiota profile as the golden standard for NEC cases. Through statistical tests, sensitivity, specificity and cut-off of selected protein levels would be assessed as prototype of diagnostic biomarkers in establishing NEC.

Sample size in this study was calculated by ANOVA repeated measure statistical analysis with a significance level of 0.05 and study power of 0.8. From the calculation, the subject needed is 10 patients for each group (total 30 subjects). The basic characteristics of the patient will be analyzed descriptively. All parameter data will be analyzed statistically by Statistical Product and Service Solution (SPSS) 20, preceded by normality test and homogeneity test. The study analysis will be sensitivity, specificity and cut-off of selected protein levels would be assessed as prototype of diagnostic biomarkers in establishing NEC. Further bivariate and multivariate analysis would be performed. Data transformation will be performed if needed in case of outlier data or out-of-range results.

ELIGIBILITY:
Inclusion Criteria of Subjects:

* Premature neonates with 28-34 weeks' gestational age
* Admitted in Perinatology Unit, Saiful Anwar General Hospital, Malang
* Parents/guardians have agreed and signed the informed consent of the study
* Neonates receive nutrition from breast milk or breast milk predominance
* NEC was diagnosed using Bell's modification criteria.

Inclusion Criteria of Control:

* Premature neonates with 28-34 weeks' gestational age, admitted in Perinatology Unit, Saiful Anwar General Hospital, Malang. Parents/guardians have agreed and signed the informed consent of the study. Neonates receive nutrition from breast milk or breast milk predominance.
* Term neonates with 37-42 weeks' gestational age, admitted in Perinatology Unit, Saiful Anwar General Hospital, Malang. Parents/guardians have agreed and signed the informed consent of the study. Neonates receive nutrition from breast milk or breast milk predominance.

Exclusion Criteria:

* Treated neonates who died during the study before the diagnosis of NEC was established
* Neonates whom require surgery during the study
* Parents/guardians stated that they were not willing to participate in the study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The target population of this study are neonates that would be categorized into three groups, i.e. preterm neonates with NEC, without NEC, and healthy term infants. The subjects are recruited from Perinatology Unit, Saiful Anwar General Hospital from March-May 2022.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change of Urinary Claudin-2 Concentration | Day-5 and Day-7 of age
  Concentrations of claudin-2 protein on Day-5 and Day-7 identified in the urine of neonates with necrotizing enterocolitis (NEC), stated numerically in ng/ml.
Change of Urinary Caveolin-1 Concentration | Day-5 and Day-7 of age
  Concentrations of caveolin-1 protein on Day-5 and Day-7 identified in the urine of neonates with necrotizing enterocolitis (NEC), stated numerically in pg/ml.
Change of Urinary EGF Concentration | Day-5 and Day-7 of age
  Concentrations of EGF protein on Day-5 and Day-7 identified in the urine of neonates with necrotizing enterocolitis (NEC), stated numerically in pg/ml.
Bell's stage of NEC | Day-1 (Baseline)
  Bell's stage of NEC are categorized into stage IIa, IIb, IIIa, and IIIb.

SECONDARY OUTCOMES:
Change of fecal microbiota profile | Day-5 and Day-7 of age
  Ratio copy number of DNA/ml feces for Proteobacteria:Firmicutes-Bacteroidetes, measured consecutively.
Change of Urinary Normalized Creatinine Level | Day-5 and Day-7 of age
  This creatinine concentration is used to normalize urinary claudin-2, caveolin-1, or EGF concentrations for ELISA.
Serum TGF-β Concentration | Day-1 (Baseline)
  Pre-existing study of TGF-β Concentration in preterm with NEC.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta IRV Corebime, M.D.(Paed), Principal Investigator — Saiful Anwar General Hospital
Locations (1):
- Saiful Anwar General Hospital, Malang, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The research team would like to discuss to what extent and the criteria of individual participant data that will be shared related to Statistical Analysis Plan, Informed Consent Form and/or Clinical Study Report.